CLINICAL TRIAL: NCT04531371
Title: Magnesium Sulphate vs Dexmedetomidine in Prevention of Emergence Agitation in Adults After Nasal Surgeries.
Brief Title: Magnesium Sulphate, Dexemeditomedine and Emergency Agitation
Acronym: agitation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ossama Hamdy Salman, clinical professor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ossamahamdyresearcher6
Record Dates: First submitted 2020-08-23; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Confusion
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dexemedetomidine (Experimental): dexemedetomidine was administered intravenously after induction of general anesthesia.
  Interventions: Drug: Dexmedetomidine injection
- magnesium sulphage (Active Comparator): magnesium sulphate was infused through out the surgery after induction of general anaesthesia.
  Interventions: Drug: Dexmedetomidine injection
- saline (Placebo Comparator): nothing was given just saline during the operation.
  Interventions: Drug: Dexmedetomidine injection

INTERVENTIONS:
Drug: Dexmedetomidine injection — post surgical agitation prophylaxis
  Other Names: dexemedetomidine

SUMMARY:
Emergence agitation is a postanesthetic phenomenon that develops in the early phase of general anesthesia recovery, and is characterized by agitation, confusion, disorientation, and possible violent behavior. Though agitation is observed more frequently in pediatric patients, the incidence in adults has been reported at 4.7% or 21.3%. Emergence agitation can lead to serious consequences such as self-extubation, removal of catheters, hemorrhage, and even severe injuries from falling out of the bed. Furthermore, it may increase the demand on human resources and cause medical staff injuries.

DETAILED DESCRIPTION:
Postoperative agitation (POA) although short-lived is potentially harmful to the patient and the recovery staff. In the postoperative care unit, an agitated patient requires more nurses to control his abnormal movement and apply restrains that could result in bruises of his extremities. In the postoperative care unit, we noticed that agitated patients remove venous and arterial catheters, nasal packs, oxygen masks and endotracheal tubes leading to bleeding and hypoxia.

Post-operative agitation is a well-documented phenomenon in children recovering from sevoflurane anesthesia. However, in adults, few reports have highlighted the occurrence of this phenomenon. The exact trigger for this complication remains to be determined, however, many factors play a crucial role in revealing POA. While an alert, calm patient is the ideal recovery outcome, the occurrence of excitation, excessive motor movements and unexplained sounds is not an uncommon scenario following nasal surgery in adults. Several factors have been incriminated to provoke agitations in adults; pain, hypoxia, type of operation, too rapid emergence from anesthesia, sedatives like benzodiazepines.

Post-operative agitation following nasal surgery The incidence of postoperative agitation following nasal surgery is relatively high. The exact mechanism is Unknown. However, some studies reported that the occurrence of POA could be as high as 55.4% and the presence of nasal pack is likely to be the main trigger of agitation. Other experiments reported an incidence of 68% following nasal surgery. We highlighted several factors that may increase the prevalence of POA; Male gender, young age, smoking, postoperative pain and premedication with atropine and Phenergan. Yu et al., 2005 reported a 55% incidence of POA after nasal surgery. They demonstrated that Doxapram administration, pain, and presence of a tracheal tube and or a urinary catheter appear to be the most important causes of postoperative agitation. Similarly, pain, urinary catheters, and tracheal tubes were also reported by Kim et al., 2004as risk factors for POA following nasal surgery. The presence of nasal pack as a trigger to POA remains debatable.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Aged 20-40 years.
* With American Society of Anesthesiologists (ASA) physical status I or II.
* Nonsmokers.
* BMI less than or equal to 30.
* Elective nasal surgery under general anesthesia in which nasal packing on each side was used postoperatively.

Exclusion Criteria:

* Patients with history of uncontrolled hypertension.
* Patients with ischemic or valvular heart disease.
* Patients use MAO inhibitors or adrenergic block.
* Cognitive impairment.
* Patients taking antipsychotics.
* Renal insufficiency or liver impairment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
post operative emergence agitation | an hour
  in post anesthetic recovery unit

CONTACTS AND LOCATIONS:
Overall Officials: Gad S Gad, MD, Study Director — South Valley University
Locations (1):
- South Valley University, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Yes